CLINICAL TRIAL: NCT00377520
Title: A Phase II Evaluation of Pemetrexed in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: A Trial for Patients With Advanced/Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8368; H3E-US-JMGT
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2009-08-24 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Neoplasms; Neoplasms by Site; Urogenital Neoplasms; Genital Neoplasms, Female; Uterine Neoplasms; Endometrial Neoplasms; Cancer of Endometrium; Endometrial Cancer; Cancer of the Endometrium; Endometrium Cancer; Neoplasms, Endometrial
MeSH Terms: conditions — Neoplasms; Neoplasms by Site; Urogenital Neoplasms; Genital Neoplasms, Female; Uterine Neoplasms; Endometrial Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 900 mg/m2, intravenous (IV), every 21 days, until disease progression
  Other Names: LY231514; Alimta

SUMMARY:
The intent of this protocol is to screen a new agent for activity in patients with advanced or recurrent endometrial carcinoma. This phase II trial is studying how well pemetrexed disodium works in treating patients with advanced or recurrent endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial adenocarcinoma, which is refractory to curative therapy or established treatments.
* Patients must have measurable disease.
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma.
* Patients must have signed an approved informed consent.
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception during the study and for at least 3 months following the last dose of Pemetrexed.
* Patients must discontinue nonsteroidal anti-inflammatory (NSAIDs) medications 2-5 days prior to and for 1-2 days after receiving Pemetrexed, depending on the half-life of the NSAIDs treatment.
* Patients must agree to this schedule in conjunction with every dose of Pemetrexed.
* Patients must receive 350-1000 mcg of folic acid (e.g. one prenatal vitamin) starting 7 days prior to the first treatment with Pemetrexed.
* Patients must be able to ingest 350-1000 mcg of folic acid daily until 3 weeks after the last dose of Pemetrexed.
* Patients must receive 4 mg Dexamethasone by mouth twice daily, 1 day prior to the dose, the day of and the day after every dose of Pemetrexed.
* Patients must receive a 1000 mcg vitamin B12 injection 7 days prior to receiving the first treatment with Pemetrexed.
* Patients must agree to receive 1000 mcg vitamin B12 injection every 9 weeks until 3 weeks after the last dose of Pemetrexed.

Exclusion Criteria:

* Patients who have had prior therapy with Pemetrexed
* Patients who have received radiation to more than 25% of marrow bearing areas

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, Study Chair — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group 215-854-0770, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed
Started | 27
Completed | 26 (Completed means the patient was evaluable for response.)
Not Completed | 1
Not completed — Ineligible (Prior radiation) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 26
Age, Customized [Number; unit: participants]
  40-49 years | 3
  50-59 years | 6
  60-69 years | 10
  >69 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 22
  Black | 3
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
Grade (Histology) [Number; unit: participants] — Assesses the extent to which cancer cells are similar in appearance and function to healthy cells of the same tissue type. Grades range from 1 (least aggressive and best prognosis) to 4 (most aggressive and worst prognosis).
  participants
    G1 - Well-Differentiated | 5
    G2 - Moderately Differentiated | 8
    G3 - Poorly Differentiated | 13
Gynecologic Oncology Group (GOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully active | 14
    1 - Ambulatory, Restricted Strenuous Activity | 12
Prior Treatment [Number; unit: participants] — Participants could have more than one type of prior treatment (radiotherapy and/or chemotherapy).
  participants
    Prior Chemotherapy | 26
    No Prior Chemotherapy | 0
    Prior Radiotherapy | 12
    No Prior Radiotherapy | 14

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment. Complete response (CR) = disappearance of all target lesions; Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions; Stable disease (SD) = small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (up to 24 months)
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 26
participants
  Completed Response | 0
  Partial Response | 1
  Stable Disease | 12
  Progressive Disease | 11
  Inevaluable | 2

2. Secondary Outcome: Number of Participants With Adverse Events by Grade (Measures of Toxicity)
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) for defining and grading specific adverse events. A grading (severity) scale is provided for each adverse event term. Grades range from 0 (none) to 5 (death). The worst grade event per cycle is reported.
Time Frame: every 21-day cycle (up to 24 months)
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 26
participants
  Leukopenia - Grade 1 | 3
  Leukopenia - Grade 2 | 4
  Leukopenia - Grade 3 | 8
  Leukopenia - Grade 4 | 2
  Thrombocytopenia - Grade 1 | 7
  Thrombocytopenia - Grade 2 | 1
  Thrombocytopenia - Grade 3 | 4
  Thrombocytopenia - Grade 4 | 0
  Neutropenia - Grade 1 | 2
  Neutropenia - Grade 2 | 3
  Neutropenia - Grade 3 | 9
  Neutropenia - Grade 4 | 3
  Anemia - Grade 1 | 9
  Anemia - Grade 2 | 11
  Anemia - Grade 3 | 5
  Anemia - Grade 4 | 0
  Coagulation - Grade 1 | 0
  Coagulation - Grade 2 | 0
  Coagulation - Grade 3 | 1
  Coagulation - Grade 4 | 0
  Nausea/vomiting - Grade 1 | 5
  Nausea/vomiting - Grade 2 | 2
  Nausea/vomiting - Grade 3 | 2
  Nausea/vomiting - Grade 4 | 0
  Gastrointestinal - Grade 1 | 6
  Gastrointestinal - Grade 2 | 6
  Gastrointestinal - Grade 3 | 3
  Gastrointestinal - Grade 4 | 0
  Alopecia - Grade 1 | 1
  Alopecia - Grade 2 | 0
  Dermatologic - Grade 1 | 4
  Dermatologic - Grade 2 | 2
  Dermatologic - Grade 3 | 1
  Dermatologic - Grade 4 | 0
  Alkaline phosphatase - Grade 1 | 4
  Alkaline phosphatase - Grade 2 | 0
  Alkaline phosphatase - Grade 3 | 0
  Alkaline phosphatase - Grade 4 | 0
  Serum glutamic-oxaloacetic transaminase - Grade 1 | 3
  Serum glutamic-oxaloacetic transaminase - Grade 2 | 0
  Serum glutamic-oxaloacetic transaminase - Grade 3 | 0
  Serum glutamic-oxaloacetic transaminase - Grade 4 | 0
  Neurologic - Grade 1 | 6
  Neurologic - Grade 2 | 3
  Neurologic - Grade 3 | 0
  Neurologic - Grade 4 | 1
  Infection - Grade 1 | 0
  Infection - Grade 2 | 4
  Infection - Grade 3 | 2
  Infection - Grade 4 | 0
  Pulmonary - Grade 1 | 2
  Pulmonary - Grade 2 | 0
  Pulmonary - Grade 3 | 0
  Pulmonary - Grade 4 | 0
  Metabolic - Grade 1 | 7
  Metabolic - Grade 2 | 1
  Metabolic - Grade 3 | 0
  Metabolic - Grade 4 | 0
  Lymphatics - Grade 1 | 3
  Lymphatics - Grade 2 | 0
  Lymphatics - Grade 3 | 1
  Lymphatics - Grade 4 | 0
  Pain - Grade 1 | 3
  Pain - Grade 2 | 2
  Pain - Grade 3 | 3
  Pain - Grade 4 | 0
  Constitutional - Grade 1 | 4
  Constitutional - Grade 2 | 8
  Constitutional - Grade 3 | 5
  Constitutional - Grade 4 | 0
  Renal - Grade 1 | 1
  Renal - Grade 2 | 0
  Renal - Grade 3 | 0
  Renal - Grade 4 | 0
  Musculoskeletal - Grade 1 | 1
  Musculoskeletal - Grade 2 | 1
  Musculoskeletal - Grade 3 | 0
  Musculoskeletal - Grade 4 | 0
  Ocular - Grade 1 | 2
  Ocular - Grade 2 | 1
  Ocular - Grade 3 | 0
  Ocular - Grade 4 | 0
  Cardiovascular - Grade 1 | 1
  Cardiovascular - Grade 2 | 1
  Cardiovascular - Grade 3 | 0
  Cardiovascular - Grade 4 | 0
  Vascular - Grade 1 | 0
  Vascular - Grade 2 | 0
  Vascular - Grade 3 | 1
  Vascular - Grade 4 | 0
  Endocrine - Grade 1 | 0
  Endocrine - Grade 2 | 1
  Endocrine - Grade 3 | 0
  Endocrine - Grade 4 | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=26)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed (N=26)
Anemia (Blood and lymphatic system disorders) | 25
Leukopenia (Blood and lymphatic system disorders) | 17
Lymphatics (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Cardiovascular (Cardiac disorders) | 2
Ocular (Eye disorders) | 3
Gastrointestinal (Gastrointestinal disorders) | 15
Nausea/vomiting (Gastrointestinal disorders) | 9
Constitutional (General disorders) | 17
Pain (General disorders) | 8
Infection (Infections and infestations) | 6
Alkaline phosphatase (Investigations) | 4
Serum glutamic-oxaloacetic transaminase (Investigations) | 3
Metabolic (Metabolism and nutrition disorders) | 8
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2
Neurologic (Nervous system disorders) | 10
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2
Dermatologic (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days